CLINICAL TRIAL: NCT07037342
Title: Immediate Effect of Acupuncture Versus Electroacupuncture on Explosive Force Production of Quadriceps Muscle in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Rowan Mohamed Raga, principle investigator : rowan mohamed raga, Egyptian Chinese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.RCT/012/004967
Record Dates: First submitted 2024-04-04; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: acupuncture; electroacupuncture; explosive force

STUDY DESIGN:
Intervention Model Description: acupuuncture and electroacupuncture
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual acupuncture (Experimental): 22 patients will receive manual acupuncture on acupoint for 20 minutes
  Interventions: Other: Manual acupuncture
- Electro acupuncture (Experimental): 22 patients will receive electro acupuncture on acupoint for 20 minutes
  Interventions: Other: Electro acupuncture
- Sham acupuncture (Sham Comparator): 22 subjects will receive sham acupuncture for 20 minutes
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Manual acupuncture — Manual acupuncture on acupoint (ST32, ST34, ST36, SP10) the needles will be inserted perpendicularly for 20 minutes.
  Arms: Manual acupuncture
Other: Electro acupuncture — Electro acupuncture on acupoint (ST32, ST34, ST36, and SP10) for 20 minutes.
  Arms: Electro acupuncture
Other: Sham acupuncture — Is a needle insertion at wrong points or non-points (locations that are not known acupuncture points)
  Arms: Sham acupuncture

SUMMARY:
The study aims to compare the immediate effects of manual needle acupuncture and electroacupuncture on the explosive force production of quadriceps in asymptomatic subjects. The hypothesis is that there will be no statistically significant difference between manual acupuncture and electroacupuncture on explosive force production.

DETAILED DESCRIPTION:
the significance of the study lies in the importance of explosive force in muscular performance, and previous research suggests that acupuncture may induce Post-activation potentiation (PAP) and improve muscle strength. However, empirical data on the immediate effects of acupuncture on explosive force production are lacking.The study will involve 66 young asymptomatic subjects divided into three groups: manual acupuncture, electroacupuncture, and sham acupuncture. Explosive force will be measured using an isokinetic device immediately after acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be asymptomatic from both genders.
* Right leg dominant .
* Age between 18 to 23.
* Body mass index ˂ 25 kg/m^2.
* Normal daily life activities.

Exclusion Criteria:

* Needles phobia.
* Under supervision of other heath practitioner.
* Involved in regular strength training during 6 months prior to the study.
* Impaired sensation or any neurological/ musculoskeletal disorder.
* Pregnant females.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Explosive force | up to twenty minutes
  Humac Norm Isokinetic dynamometer will be used for measuring explosive force performance

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Chinese University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No